CLINICAL TRIAL: NCT05171283
Title: Oat Fiber and Cardiovascular Risk Reduction: A Systematic Review and Meta-analysis of Randomized Controlled Trials
Brief Title: Meta-analysis of Oat Fiber and Cardiovascular Risk Reduction
Status: Active, not recruiting | Type: Observational
Sponsor: University of Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Quaker Oats Centre of Excellence, Quaker (Unknown)
Responsible Party: Principal Investigator, John Sievenpiper, Associate Professor, University of Toronto
Other Study IDs: CIHR - Oats and CVD Risk
Record Dates: First submitted 2021-11-18; First posted 2021-12-28 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Cardiovascular Diseases; Coronary Heart Disease
Keywords: Oat; Oat fibre; beta-glucan; Avena sativa; Systematic reviews and meta-analysis; Clinical practice guidelines; Controlled trials; Cardiovascular disease; Coronary heart disease; 10-year cardiovascular risk score
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Gyrate Atrophy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Oats or Oat Fibre — Interventions that contain whole grain oats or oat beta-glucan.

SUMMARY:
Oat fibre has been shown to lower cholesterol and may have cardioprotective effects. However, whether this translates to actual cardiovascular risk reduction is unclear, as there is a lack of controlled human trials. To address this uncertainty, the investigator proposes to use established cardiovascular disease risk scores, such as those recommended by the Canadian Cardiovascular Society and other clinical practice groups, to create composite risk scores in assessing future risk. The data on oat fibre will be collected through a systematic review of controlled trials, composite cardiovascular risk scores will be calculated for each eligible study, and meta-analyses will be conducted to assess the overall effect. The findings generated by this proposed knowledge synthesis will help improve the health of consumers through informing evidence-based guidelines and improving health outcomes by educating healthcare providers and patients, stimulating industry innovation, and guiding future research design.

DETAILED DESCRIPTION:
Background: Although oat beta-glucan has an approved health claim for cholesterol-lowering in Canada, US, and Europe, it is unclear whether this effect translates into lower cardiovascular disease risk. There is a well-established causal link between LDL-C and cardiovascular disease based on the results of pharmacological interventions that target different LDL-C- lowering mechanisms and mendelian randomization studies. However, there are no randomized controlled trials of the effect of whole grain oats or oat beta-glucan on cardiovascular outcomes and the few prospective cohort studies that have assessed the relation of whole grain oats with cardiovascular outcomes have failed to show a reliable protective association.

One way to confirm the cardiovascular benefit of whole grain oats and oat beta-glucan would be to use an established 10-year cardiovascular disease risk score such as the modified Framingham Risk Score (FRS) (recommended by the Canadian Cardiovascular Society [CCS]), the American College of Cardiology/American Heart Association (ACC/AHA) ASCVD risk estimator (recommended by the ACC/AHA) or Systemic Coronary Risk Estimation (SCORE) (recommended by the European Society of Cardiology [ESC] and European Atherosclerosis Society [EAS]). These scores are composites of cardiovascular risk factors in which cholesterol and blood pressure carry important weight. There are numerous systematic reviews and meta-analyses of randomized trials showing a benefit of whole grain oats and oat beta-glucan for cholesterol and blood pressure. The investigators propose a novel approach to leverage these benefits to detect an overall reduction in 10-year cardiovascular disease by these scores.

Need for proposed research: High quality systematic reviews and meta-analyses of randomized controlled trials represent the highest level of evidence to support dietary guidelines and public health policy development. As dietary guidelines and public health policy have shifted toward food and dietary-pattern based recommendations, there is a need for systematic reviews and meta-analyses on the effect of oats and oat beta-glucan on cardiovascular risk.

Objective: To improve evidence-based guidance for clinical practice guidelines for nutrition therapy and public health policy development, the investigators will conduct a systematic review and meta-analysis of the effects of whole grain oats and oat beta-glucan on 10-year cardiovascular disease risk using (1) the modified Framingham Risk Score, (2) the ASCVD risk estimator, and (3) the SCORE.

Design: The systematic review and meta-analysis will be conducted according to the Cochrane Handbook for Systematic Reviews of Interventions and reported according to the Preferred Reporting Items for Systematic Reviews and Meta-Analyses (PRISMA).

Data sources: MEDLINE, EMBASE, and The Cochrane Central Register of Controlled Trials (Clinical Trials; CENTRAL) will be searched using appropriate search terms supplemented by manual searches of references of included studies.

Study selection: The investigators will include randomized controlled trials of ≥3-weeks in adults of all health backgrounds assessing the effect of oat beta-glucan compared with a suitable non-beta-glucan control on 10-year cardiovascular risk calculated by the 3 cardiovascular risk scores which will require data on a combination of blood lipids (total-cholesterol and HDL-cholesterol) and systolic blood pressure (for calculation of the 3 scores). Studies that are not conducted in humans, not randomized, have an acute feeding design (<3 weeks), lack a suitable control (non-isocaloric, contain beta-glucan) and/or do not report viable endpoint data will not be included.

Data extraction: Two or more investigators will independently extract relevant data and assess risk of bias using the Cochrane Risk of Bias Tool. All disagreements will be resolved by consensus.. Authors will be contacted for additional information and standard computations and imputations will be used to derive missing variance data.

Outcomes: The primary outcome will be the between treatment change in the modified Framingham Risk Score (FRS) to estimate 10-year risk of cardiovascular disease (https://www.ccs.ca/images/Guidelines/Tools_and_Calculators_En/FRS_eng_2017_fnl1.pdf). Secondary outcomes include the between treatment change in the American College of Cardiology/American Heart Association (ACC/AHA) ASCVD risk estimator (https://tools.acc.org/ascvd-risk-estimator-plus/#!/calculate/estimate/) to estimate the 10-year risk of atherosclerotic cardiovascular disease (ASCVD) and in the Systemic Coronary Risk Estimation (SCORE) (https://www.escardio.org/Education/Practice-Tools/CVD-prevention-toolbox/SCORE-Risk-Charts) derived by the European Society of Cardiology to estimate 10-year risk of cardiovascular disease. Additional outcomes include between treatment changes in the modifiable components of all the scores: total-cholesterol, HDL-cholesterol, and systolic blood pressure.

Data synthesis: Separate pooled analyses will be conducted for each cardiovascular risk score using the Generic Inverse Variance method. Random-effects models will be used even in the absence of statistically significant between-study heterogeneity, as this yield more conservative summary effect estimates in the presence of residual heterogeneity. Exceptions will be made for the use of fixed-effects models where there is <5 included trials irrespective of heterogeneity or small trials are being pooled with larger more precise trials in the absence of statistically significant heterogeneity. Paired analyses will be applied to all crossover trials. Heterogeneity will be tested by Cochran's Q statistic and quantified by the I2 statistic. To explore sources of heterogeneity, the investigators will conduct sensitivity analyses, in which each study is systematically removed. If there are ≥10 studies, then the investigators will also explore sources of heterogeneity by a priori subgroup analyses by study design (parallel or crossover), follow-up duration (<12 weeks or ≥12 weeks), comparator diet, baseline risk, risk of bias and background health status. Significant unexplained heterogeneity will be investigated by additional post hoc subgroup analyses by age (<18y vs ≥18y), energy balance (neutral, negative or positive), feeding control (metabolic, supplemented, dietary advice, ad libitum), and funding. Meta-regression analyses will assess the significance of categorical and continuous subgroups analyses. Linear dose-response analyses will be assessed using continuous meta-regression analyses. Non-linear dose-response association will be assessed using a two-stage multivariate random-effects method with restricted cubic splines with three knots. When ≥10 studies are available, publication bias will be investigated by inspection of funnel plots and formal testing using the Egger's and Begg's tests. If publication bias is suspected, then the investigators will attempt to adjust for funnel plot asymmetry by imputing the missing study data using the Duval and Tweedie trim and fill method.

Evidence assessment: The strength of the evidence for each outcome will be assessed using the Grading of Recommendations Assessment, Development and Evaluation (GRADE).

Knowledge translation plan: The results will be disseminated through interactive presentations at local, national, and international scientific meetings and publication in high impact factor journals. Target audiences will include the public health and scientific communities with interest in nutrition, diabetes, obesity, and cardiovascular disease. Feedback will be incorporated and used to improve the public health message and key areas for future research will be defined. Applicant/Co-applicant Decision Makers will network among opinion leaders to increase awareness and participate directly as committee members in the development of future guidelines.

SIGNIFICANCE The proposed project will aid in knowledge translation related to the role of oats in cardiovascular risk reduction strengthening the evidence-base for guidelines development in the U.S., Canada, Europe, and beyond and improving health outcomes, by educating healthcare providers and patients, stimulating industry innovation, and guiding future research design.

ELIGIBILITY:
Inclusion Criteria:

* Dietary trials in humans
* Randomized treatment allocation
* ≥3 weeks
* Intervention with oats or oat beta-glucan
* Suitable control (i.e. isocaloric diet that is not vegetarian or vegan)
* Ascertainment of viable outcome data for cardiovascular risk calculations

Exclusion Criteria:

* Non-human studies
* Non-randomized treatment allocation
* <3 weeks
* No intervention of oats or oat beta-glucan
* Lack of a suitable control (i.e. non-isocaloric)
* No viable endpoint data

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Any population type.
Sampling Method: Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Framingham Risk Score (FRS) | >= 3-weeks
  Framingham Risk Score (FRS) calculates 10-year cardiovascular risk using the Cox formula which includes age, sex, total cholesterol, HDL-cholesterol, systolic blood pressure, blood pressure medication use, diabetes status, smoking status; minimum score 0%, maximum score 100% where higher score indicates higher risk of 10-year risk of cardiovascular disease

SECONDARY OUTCOMES:
ACC/AHA ASCVD risk estimator | >= 3-weeks
  American College of Cardiology/American Heart Association (ACC/AHA) risk estimator calculates 10-year risk of atherosclerotic cardiovascular disease (ASCVD) using a formula which includes age, sex, race, total cholesterol, HDL-cholesterol, systolic blood pressure, blood pressure medication use, diabetes status, smoking status; minimum score 0, maximum score 100 where higher score indicates higher risk of 10-year risk of atherosclerotic cardiovascular disease (ASCVD)
Systematic COronary Risk Evaluation (SCORE) | >= 3-weeks
  European Society of Cardiology derived "SCORE" calculates 10-year risk of cardiovascular disease using a formula which includes age, sex, country, total cholesterol, systolic blood pressure, blood pressure medication use, diabetes status, smoking status; minimum score 0, maximum score 100 where higher score indicates higher risk of 10-year risk of cardiovascular disease

OTHER OUTCOMES:
Modifiable components of the risk scores - total-cholesterol | >= 3-weeks
  total-cholesterol
Modifiable components of the risk scores - HDL-cholesterol | >= 3-weeks
  HDL-cholesterol
Modifiable components of the risk scores - systolic blood pressure | >= 3-weeks
  Systolic blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: John L Sievenpiper, PhD, MD, Principal Investigator — University of Toronto
Locations (1):
- The Toronto 3D (Diet, Digestive tract and Disease) Knowledge Synthesis and Clinical Trials Unit, Clinical Nutrition and Risk Factor Modification Centre, St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
All data will be available in the publication.

REFERENCES:
- [Background] Food Directorate Health Products and Food Branch, Health Canada Oat products and blood cholesterol lowering Bureau of Nutritional Sciences, Ottawa (2010). Available at https://www.canada.ca/en/health-canada/services/food-nutrition/food-labelling/health-claims/assessments/products-blood-cholesterol-lowering-summary-assessment-health-claim-about-products-blood-cholesterol-lowering.html
- [Background] U.S. Food & Drug Administration, Health and Human Services. Food Labeling: Health Claims; Soluble Dietary Fiber From Certain Foods and Coronary Heart Disease. 21 CFR Part 101 [Docket No. 01Q-0313]. Available at https://www.gpo.gov/fdsys/pkg/FR-2002-10-02/pdf/02-25067.pdf
- [Background] EFSA Panel on Dietetic Products, Nutrition and Allergies (NDA) Scientific Opinion on the substantiation of a health claim related to oat beta-glucan and lowering blood cholesterol and reduced risk of (coronary) heart disease pursuant to Article 14 of Regulation (EC) No 1924/2006 EFSA J, 8 (12) (2010), p. 1885, 10.2903/j.efsa.2010.1885 Available at www.efsa.europa.eu/efsajournal.htm
- [Background] Ference BA, Cannon CP, Landmesser U, Luscher TF, Catapano AL, Ray KK. Reduction of low density lipoprotein-cholesterol and cardiovascular events with proprotein convertase subtilisin-kexin type 9 (PCSK9) inhibitors and statins: an analysis of FOURIER, SPIRE, and the Cholesterol Treatment Trialists Collaboration. Eur Heart J. 2018 Jul 14;39(27):2540-2545. doi: 10.1093/eurheartj/ehx450. No abstract available. PMID 29020411
- [Background] Ference BA, Robinson JG, Brook RD, Catapano AL, Chapman MJ, Neff DR, Voros S, Giugliano RP, Davey Smith G, Fazio S, Sabatine MS. Variation in PCSK9 and HMGCR and Risk of Cardiovascular Disease and Diabetes. N Engl J Med. 2016 Dec 1;375(22):2144-2153. doi: 10.1056/NEJMoa1604304. PMID 27959767
- [Background] Helnaes A, Kyro C, Andersen I, Lacoppidan S, Overvad K, Christensen J, Tjonneland A, Olsen A. Intake of whole grains is associated with lower risk of myocardial infarction: the Danish Diet, Cancer and Health Cohort. Am J Clin Nutr. 2016 Apr;103(4):999-1007. doi: 10.3945/ajcn.115.124271. Epub 2016 Feb 17. PMID 26888710
- [Background] Johnsen NF, Frederiksen K, Christensen J, Skeie G, Lund E, Landberg R, Johansson I, Nilsson LM, Halkjaer J, Olsen A, Overvad K, Tjonneland A. Whole-grain products and whole-grain types are associated with lower all-cause and cause-specific mortality in the Scandinavian HELGA cohort. Br J Nutr. 2015 Aug 28;114(4):608-23. doi: 10.1017/S0007114515001701. Epub 2015 Jul 23. PMID 26201847
- [Background] Juan J, Liu G, Willett WC, Hu FB, Rexrode KM, Sun Q. Whole Grain Consumption and Risk of Ischemic Stroke: Results From 2 Prospective Cohort Studies. Stroke. 2017 Dec;48(12):3203-3209. doi: 10.1161/STROKEAHA.117.018979. Epub 2017 Nov 10. PMID 29127271
- [Background] Goff DC Jr, Lloyd-Jones DM, Bennett G, Coady S, D'Agostino RB Sr, Gibbons R, Greenland P, Lackland DT, Levy D, O'Donnell CJ, Robinson JG, Schwartz JS, Shero ST, Smith SC Jr, Sorlie P, Stone NJ, Wilson PWF. 2013 ACC/AHA guideline on the assessment of cardiovascular risk: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines. J Am Coll Cardiol. 2014 Jul 1;63(25 Pt B):2935-2959. doi: 10.1016/j.jacc.2013.11.005. Epub 2013 Nov 12. No abstract available. PMID 24239921
- [Background] Anderson TJ, Gregoire J, Pearson GJ, Barry AR, Couture P, Dawes M, Francis GA, Genest J Jr, Grover S, Gupta M, Hegele RA, Lau DC, Leiter LA, Lonn E, Mancini GB, McPherson R, Ngui D, Poirier P, Sievenpiper JL, Stone JA, Thanassoulis G, Ward R. 2016 Canadian Cardiovascular Society Guidelines for the Management of Dyslipidemia for the Prevention of Cardiovascular Disease in the Adult. Can J Cardiol. 2016 Nov;32(11):1263-1282. doi: 10.1016/j.cjca.2016.07.510. Epub 2016 Jul 25. PMID 27712954
- [Background] Catapano AL, Graham I, De Backer G, Wiklund O, Chapman MJ, Drexel H, Hoes AW, Jennings CS, Landmesser U, Pedersen TR, Reiner Z, Riccardi G, Taskinen MR, Tokgozoglu L, Monique Verschuren WM, Vlachopoulos C, Wood DA, Luis Zamorano J; Additional Contributor; Cooney MT. 2016 ESC/EAS Guidelines for the Management of Dyslipidaemias. Rev Esp Cardiol (Engl Ed). 2017 Feb;70(2):115. doi: 10.1016/j.rec.2017.01.002. No abstract available. English, Spanish. PMID 29389351
- [Background] Ho HV, Sievenpiper JL, Zurbau A, Blanco Mejia S, Jovanovski E, Au-Yeung F, Jenkins AL, Vuksan V. The effect of oat beta-glucan on LDL-cholesterol, non-HDL-cholesterol and apoB for CVD risk reduction: a systematic review and meta-analysis of randomised-controlled trials. Br J Nutr. 2016 Oct;116(8):1369-1382. doi: 10.1017/S000711451600341X. Epub 2016 Oct 11. PMID 27724985
- [Background] Hollaender PL, Ross AB, Kristensen M. Whole-grain and blood lipid changes in apparently healthy adults: a systematic review and meta-analysis of randomized controlled studies. Am J Clin Nutr. 2015 Sep;102(3):556-72. doi: 10.3945/ajcn.115.109165. Epub 2015 Aug 12. PMID 26269373
- [Background] Khan K, Jovanovski E, Ho HVT, Marques ACR, Zurbau A, Mejia SB, Sievenpiper JL, Vuksan V. The effect of viscous soluble fiber on blood pressure: A systematic review and meta-analysis of randomized controlled trials. Nutr Metab Cardiovasc Dis. 2018 Jan;28(1):3-13. doi: 10.1016/j.numecd.2017.09.007. Epub 2017 Oct 7. PMID 29153856
- [Background] Higgins JPT, Greens S (editors). Cochrane Handbook for Systematic Reviews of Interventions Version 5.1.0 [updated March 2011]. The Cochrane Collaboration, 2011. Available from www.cochrane-handbook.org.
- [Background] Moher D, Liberati A, Tetzlaff J, Altman DG; PRISMA Group. Preferred reporting items for systematic reviews and meta-analyses: the PRISMA statement. J Clin Epidemiol. 2009 Oct;62(10):1006-12. doi: 10.1016/j.jclinepi.2009.06.005. Epub 2009 Jul 23. No abstract available. PMID 19631508
- [Background] Elbourne DR, Altman DG, Higgins JP, Curtin F, Worthington HV, Vail A. Meta-analyses involving cross-over trials: methodological issues. Int J Epidemiol. 2002 Feb;31(1):140-9. doi: 10.1093/ije/31.1.140. PMID 11914310
- [Background] Graham ID, Logan J. Innovations in knowledge transfer and continuity of care. Can J Nurs Res. 2004 Jun;36(2):89-103. PMID 15369167